CLINICAL TRIAL: NCT05901311
Title: A Phase I, Open-label, Two-part Study of the Absorption, Metabolism, Excretion, and the Absolute Bioavailability of [14C]-LY3537982 in Healthy Adult Subjects
Brief Title: A Study of [14C]-LY3537982 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-RAS-23003; J3M-OX-JZQE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [¹⁴C]-LY3537982 (Part 1) (Experimental): Single dose of [¹⁴C]-LY3537982 administered orally.
  Interventions: Drug: [¹⁴C]-LY3537982
- [¹⁴C]-LY3537982 + LY3537982 (Part 2) (Experimental): Single dose of LY3537982 administered orally followed by [¹⁴C]-LY3537982 administered intravenously (IV).
  Interventions: Drug: LY3537982; Drug: [¹⁴C]-LY3537982

INTERVENTIONS:
Drug: LY3537982 — Administered orally.
  Other Names: Olomorasib
  Arms: [¹⁴C]-LY3537982 + LY3537982 (Part 2)
Drug: [¹⁴C]-LY3537982 — Administered orally.
  Arms: [¹⁴C]-LY3537982 (Part 1)
Drug: [¹⁴C]-LY3537982 — Administered IV.
  Arms: [¹⁴C]-LY3537982 + LY3537982 (Part 2)

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much LY3537982 is in the bloodstream and how the body handles and eliminates LY3537982 in healthy participants. This study will involve a single dose of 14C radiolabeled LY3537982. This means that a radioactive tracer substance, C14, will be incorporated into the study drug LY3537982 to investigate the study drug and its breakdown products and to find out how much of these passes from blood into urine, feces and expired air. The study will also evaluate the safety and tolerability of LY3537982. The study will be conducted in two parts. The study will last up to 71 days and 61 days for part 1 and 2, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants in good health, determined by no clinically significant findings from medical history, physical examination as assessed by the investigator.
* Have a body mass index within the range 18.5 to 32.0 kilograms per meter squared (kg/m²)
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods.

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Fraction of Dose Excreted in Urine (Feur) | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Feur
PK: Cumulative Feur | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Cumulative Feur
PK: Fraction of Dose Excreted in Feces (Fefeces) | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Fefeces
PK: Cumulative Fefeces | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Cumulative Fefeces
PK: Fraction of Dose Excreted in Expired Air (Feair) | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Feair
PK: Absolute Bioavailability (F) of LY3537982 | Predose on day 1 up to postdose on day 9 (Part 2)
  PK: F of LY3537982

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Labcorp Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No